CLINICAL TRIAL: NCT02671734
Title: Using Media to Improve the Informed Consent Process for Youth Undergoing Pediatric Endoscopy and Their Parents
Brief Title: Improving the Informed Consent Process for Youth Undergoing Pediatric Endoscopy and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huang, Jeannie, M.D. (Individual)
Responsible Party: Principal Investigator, Jeannie Huang, MD, MPH, Associate Professor, Huang, Jeannie, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 121426
Record Dates: First submitted 2016-01-25; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Children
Keywords: endoscopy
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): Subjects in this arm received the standard consent form to read and underwent standard discussions with the procedurist prior to the procedure.
- intervention (Active Comparator): Subjects in this arm viewed a video detailing key elements of informed consent. Subjects in this arm also received the standard consent form to read and underwent standard discussions with the procedurist prior to the procedure.
  Interventions: Behavioral: video

INTERVENTIONS:
Behavioral: video — Short (2 minute 43 second), animated videos were designed addressing nature of the procedure, risks, benefits, and alternatives for upper and lower endoscopy respectively using PowToon (www.powtoon.com). Sixth grade language was used throughout the video. Videos were shown to youth and their parents on an iPad.
  Arms: intervention

SUMMARY:
The investigators employed a randomized control study design to evaluate the efficacy of a video intervention augmenting informed consent discussions in improving parental and youth informed consent comprehension.

DETAILED DESCRIPTION:
IC = informed consent

The investigators employed a randomized control study design to evaluate the efficacy of a video intervention augmenting IC discussions in improving parental and youth IC comprehension. Sample size was selected to detect a 30% improvement in comprehension scores in the intervention v. control group. The local Institutional Review Board approved the study. Informed consent and assent were obtained prior to all study procedures.

ELIGIBILITY:
Inclusion Criteria:

* For children admitted, age limits listed. Youth-parent pairs were admitted into the study.
* Had to be undergoing pediatric endoscopy.
* English speaking

Exclusion Criteria:

* None.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of Comprehension of Informed Consent Process via a scored scale | Day 1
  Structured Interview

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie Huang, MD, MPH, Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: No